CLINICAL TRIAL: NCT03235453
Title: Influence of Binary and Quaternary Rhythm in Motor Symptoms, Sleep, Failure and Quality of Living in People With Parkinson Disease: a Randomized Clinical Trial
Brief Title: Dance for People With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laboratório de Pesquisa em Lazer e Atividade Física (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 71690317700000118
Record Dates: First submitted 2017-07-28; First posted 2017-08-01 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Parkinson Disease; Quality of Life; Sleep Disorder; Gait Disorders, Neurologic; Mobility Limitation
Keywords: Parkinson; Quality of Life; Sleep Disorder; Gait Disorders; Mobility
MeSH Terms: conditions — Parkinson Disease; Sleep Wake Disorders; Gait Disorders, Neurologic; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial, two arm study (group 1 - Binary Rhythm; group 2 - Quaternary Rhythm
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binary rhythm (Experimental): Experimental: binary rhythm The randomized group for binary-rhythm intervention will receive a 12-week intervention with dance lessons. Classes will be divided into: Heating and stretching (5 minutes), main part (binary) (35 minutes) and relaxation (5 minutes).
  Interventions: Other: Binary rhythm
- Quaternary rhythm (Experimental): The randomized group for the quaternary rhythm intervention will receive a 12-week intervention with dance classes. Classes will be divided into: Heating and stretching (5 minutes), main part (quaternary rhythm) (35 minutes) and relaxation (5 minutes).
  Interventions: Other: Quaternary rhythm

INTERVENTIONS:
Other: Binary rhythm — The binary rhythm intervention will be performed using the dance modalities, Forró, Merengue and Bolero. It will occur twice a week for 12 weeks with 45 minutes of sitting.
  Other Names: Dance
  Arms: Binary rhythm
Other: Quaternary rhythm — The quaternary rhythm intervention will be performed using the modalities of dance, Tango, Salsa, Zouk. It will occur twice a week for 12 weeks with 45 minutes of sitting.
  Other Names: Dance
  Arms: Quaternary rhythm

SUMMARY:
The randomized clinical trial will aim to analyze the influence of binary and quaternary rhythm through a protocol on motor symptoms, sleep, fatigue and quality of life in individuals with Parkinson's disease. The study design with a randomized clinical trial, including individuals diagnosed with Parkinson's Disease, will be divided into two groups: 1) Control group 2) Experimental group. Cognition, balance, gait freezing, functional mobility, quality of life, sleep, daytime sleepiness and fatigue will be evaluated. Through the application of binary and quaternary rhythm protocol for a period of 12 weeks. First, the descriptive statistics (mean, standard deviation and percentage) will be used to know the data, then the normality calculation using the Kolmogorov Smirnov test will be used to choose the statistical tests. All information will be collected before and after the intervention period. For statistical analysis, use the SPSS statistical package, version 20.0. (Kolmogorov-Smirnov or Shapiro-Wilk test) for the selection of statistical tests.

DETAILED DESCRIPTION:
The project includes two protocols: (1) Dance binary rhythm and (2) Dance quaternary rhythm. Each session will last 45 minutes for each modality, twice a week, over a period of 12 weeks. Blood pressure (BP) and heart rate will be seen at the beginning and end of each class. In addition to the Effort Perception Scale - Borg Scale used to assess the intensity and / or discomfort during physical activity practice in both protocols. In both modalities of intervention, the evolution of the movements will always respect the limit of each patient. The binary rhythm protocol will be performed through forró, meringue and bolero rhythms, this type of methodology was selected, because it is a stimulating rhythm that brings harmony of the movements, being able to be associated to improvements in the mobility, balance and quality of life of the individuals who Practice it, benefiting patients directly.

The binary protocol classes will be divided into: heating (10 minutes) focused on dance styles that contemplate the binary rhythm, with walks in the marking of the musical rhythm, muscular release, breathing, movements for upper and lower limbs, always working musicality . The main part (30 minutes) will be divided into two moments, first individually so that the teacher can show and teach in a clear way the steps that will be performed then the participants will form pairs and perform the steps that were taught them. Every 5 minutes the participants will change their pair, so that everyone can have the experience of dancing with their colleagues. And to finish it will be carried out a calm return (5 minutes) to provide muscular relaxation with stretches and massages.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PD following the criteria of the brain bank of London.
* Individuals of both sexes, aged 25 years or older.
* With stable doses of the medication, in the "On" phase of the medication.

Exclusion Criteria:

* Individuals who do not complete all study steps.
* That they are not stable in doses of medication.

Ages: 25 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-30 (Estimated); Primary Completion 2017-12-30 (Estimated); Study Completion 2019-12-20 (Estimated)

PRIMARY OUTCOMES:
Balance | 10 minutes
  The Mini-BESTest test is a 14-item test that focuses on dynamic balance, specifically anticipated transitions, postural responses, sensory orientation, and dynamic gait. Each item is scored from (0-2); A score of 0 indicates that a person is unable to perform the task while a score of 2 is normal.
Gait | 10 minutes
  Freezing of Gait - FOG-Q - The score for each item ranges from zero to four, with higher scores indicating more severe freezing episodes. It presents a total score of 24, and the highest score represents a severe gait impairment
Mobility | 5 minutes
  Timed Up & Go (TUG), The TUG measures the time it takes an individual to perform some functional maneuvers, such as getting up, walking, taking a walk, and sitting down.
  A) less than 20 seconds to perform, corresponds to low risk for falls. B) from 20 to 29 seconds, at medium risk for falls. C) 30 seconds or more at high risk for falls

SECONDARY OUTCOMES:
Quality of life | 5 minutes
  The Parkinson's Disease Questionnaire - PDQ-39 Is a specific scale of evaluation of quality of life in PD, comprises 39 items that can be answered with five different response options: "never"; "On occasion"; "sometimes"; "often"; "Always" or "impossible for me". The scores on each item range from 0 (never) to 4 (always or impossible for me).
Sleep | 5 minutes
  Parkinson's Sleep Scale (PDSS)- Addresses 15 symptoms associated with sleep disorders.The maximum score for PDSS is 150 (patient is free of all symptoms)
Daytime sleepiness | 5 minutes
  The Epworth Sleepiness Scale It is a self-administered questionnaire that evaluates the probability of falling asleep in eight situations involving daily activities, The overall score ranges from 0 to 24, with scores above 10 suggesting the diagnosis of excessive daytime sleepiness
Fatigue | 5 minutes
  Fatigue Severity Scale: an instrument for evaluating the physical aspects of fatigue and its impact on the daily function of the patient. The FSS total score represents the average score of the nine articles ranging from 1 to 7, in which the higher scores indicate more severe fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Jéssica Moratelli, Principal Investigator — University of the State of Santa Catarina; Adriana CA Guimarães, PhD, Study Director — University of the State of Santa Catarina; Kettlyn Hames, Principal Investigator — University of the State of Santa Catarina

IPD SHARING:
Plan to Share IPD: No